CLINICAL TRIAL: NCT04735523
Title: Replication of the RECOVER-II Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-RE-COVER II
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Dabigatran: Exposure group
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Dabigatran dispensing claim is used as the exposure group
  Groups: Dabigatran
Drug: Warfarin — Warfarin dispensing claim is used as the reference group
  Groups: Warfarin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Market availability of dabigatran in the U.S. for treatment of deep vein thrombosis and pulmonary embolism started on April 7, 2014

* For Medicare: April 7, 2014 - December 31, 2017 (end of available data)
* For Marketscan: April 7, 2014 - December 31, 2018 (end of available data)
* For Optum: April 7, 2014 - March 31, 2020 (end of available data)

Inclusion Criteria:

* Acute deep vein thrombosis (DVT) of the leg involving proximal veins, and/or pulmonary embolism (PE) iin patients for whom at least 6 months of anticoagulant therapy is considered appropriate.
* Men and women ages 18 years or greater

Exclusion Criteria:

* PE satisfying at least one of the following criteria:

  * Haemodynamic instability
  * OR Embolectomy is indicated or performed
  * OR thrombolytic therapy is indicated or performed
  * OR suspected source of PE is other than blood clots from the legs
* Actual or anticipated use of vena cava filter
* Patients who in the investigators judgement are perceived as having an excessive risk of bleeding
* Known anaemia
* Need of anticoagulant treatment for disorders other than VTE
* Recent unstable cardiovascular disease
* Elevated AST or ALT > 3x ULN
* Liver disease expected to have any potential impact on survival (severe liver conditions)
* Severe renal impairment
* Contraindications to anticoagulant therapy (not specified)
* Recent or active major bleeding
* Recent brain, eye, or spinal cord injury or surgery
* Malignant or severe, uncontrolled hypertension
* Active infective endocarditis
* Mechanical prosthetic heart valve (recently implanted - RE-ALIGN trial)
* Women who are pregnant, nursing, or of childbearing potential who refuse to use a medically acceptable form of contraception
* Patients who have developed transaminase elevations upon exposure to ximelagatran
* Patients considered unsuitable for inclusion by the investigator

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing dabigatran to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of dabigatran to warfarin (index date). We will restrict the analyses to patients with a diagnosis of proximal DVT or PE.
Sampling Method: Non-Probability Sample
Enrollment: 5350 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
VTE and cause-specific mortality | Through study completion (a median of 84-89 days)

SECONDARY OUTCOMES:
Hospital admission for VTE | Through study completion (a median of 84-89 days)
Cause-specific mortality | Through study completion (a median of 84-89 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT04735523/Prot_001.pdf